CLINICAL TRIAL: NCT02244632
Title: An Open-label, Multiple-site, Phase I/II Dose Cohort Trial of [6R] 5,10-Methylene Tetrahydrofolate (Modufolin®) in Combination With a Fixed Dose of 5-Fluorouracil (5-FU) Alone or Together With a Fixed Dose of Oxaliplatin or Irinotecan in Patients With Stage IV Colorectal Cancer
Brief Title: Modufolin (Arfolitixorin) in Combination With 5-Fluorouracil Alone or Together With Oxaliplatin or Irinotecan in Colorectal Cancer
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Isofol Medical AB (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ISO-CC-005; 2014-001862-84 (EudraCT Number)
Record Dates: First submitted 2014-09-17; First posted 2014-09-19 (Estimated); Last update posted 2020-09-09 (Actual); Status verified 2020-09

CONDITIONS: Colorectal Neoplasm
Keywords: Colorectal cancer; Colorectal carcinoma; Colorectal tumors; Intestinal Neoplasm; Gastrointestinal Neoplasm; Gastrointestinal disease; 5,10-methylenetetrahydrofolate; Tetrahydrofolates; Therapeutic uses; Pharmacokinetics; Pharmacodynamics; Safety assessments
MeSH Terms: conditions — Colorectal Neoplasms; Intestinal Neoplasms; Gastrointestinal Neoplasms; Gastrointestinal Diseases | interventions — 5,10-methylenetetrahydrofolic acid; Fluorouracil; Oxaliplatin; Irinotecan; Bevacizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (6):
- Modufolin / Nordic FLV (Experimental): Modufolin in combination with 5-Fluorouracil only.
  Interventions: Drug: Modufolin (arfolitixorin); Drug: Fluorouracil
- Modufolin / Nordic FLOX (Experimental): Modufolin in combination with 5-Fluorouracil and Oxaliplatin according to Nordic FLOX regime
  Interventions: Drug: Modufolin (arfolitixorin); Drug: Fluorouracil; Drug: Oxaliplatin
- Modufolin / Nordic FLIRI (Experimental): Modufolin in combination with 5-Fluorouracil and Irinotecan.
  Interventions: Drug: Modufolin (arfolitixorin); Drug: Fluorouracil; Drug: Irinotecan
- MOFOX (Experimental): Modufolin in combination with 5-Fluorouracil and Oxaliplatin according to mFOLFOX-6 regime
  Interventions: Drug: Modufolin (arfolitixorin); Drug: Fluorouracil; Drug: Oxaliplatin
- MOFOX / Bevacizumab (Experimental): Modufolin in combination with 5-Fluorouracil, Oxaliplatin and Bevacizumab
  Interventions: Drug: Modufolin (arfolitixorin); Drug: Fluorouracil; Drug: Oxaliplatin; Drug: Bevacizumab
- MOFIRI (Experimental): Modufolin in combination with 5-Fluorouracil and Irinotecan
  Interventions: Drug: Modufolin (arfolitixorin); Drug: Fluorouracil; Drug: Irinotecan

INTERVENTIONS:
Drug: Modufolin (arfolitixorin) — IV injection every second week for 8 weeks.
  Other Names: [6R] 5,10-methylenetetrahydrofolate; 6R-MTHF; 6R-methylene THF; ISO-901; arfolitixorin
Drug: Fluorouracil — IV injection every second week for 8 weeks.
  Other Names: 5-FU; 5-Flourouacil; 5-Fluoro-1H,3H-pyrimidine-2,4-dione; Adrucil
Drug: Oxaliplatin — IV infusion every second week for 8 weeks.
  Other Names: Eloxatin; [(1R,2R)-cyclohexane-1,2-diamine](ethanedioato-O,O')platinum(II); Olatin; Oxamed; Oxitropic
  Arms: MOFOX; MOFOX / Bevacizumab; Modufolin / Nordic FLOX
Drug: Irinotecan — IV infusion every second week for 8 weeks.
  Other Names: (+)-(4S)-4,11-Dietyl-4-hydroxi-9-[(4-piperidinopiperidino)karbonyloxi]-1H-pyrano[3¢,4¢:6,7]indolizino[1,2-b]kinolin-3,14-(4H,12H)dion; Irinosor; Campto; Namedica
  Arms: MOFIRI; Modufolin / Nordic FLIRI
Drug: Bevacizumab — IV infusion every second week for 8 weeks.
  Other Names: Avastin
  Arms: MOFOX / Bevacizumab

SUMMARY:
The purpose is to characterise the tolerability of Modufolin (arfolitixorin) in combination with 5-FU alone, in combination with 5-FU and Oxaliplatin, in combination with 5-FU and Irinotecan and in combination with 5-FU, Oxaliplatin and Bevacizumab.

Another purpose is to investigate 4 doses of Modufolin to identify the best dose for further assessment.

DETAILED DESCRIPTION:
The study will investigate the tolerability of Modufolin at four (4) different dose levels (30 to 240 mg/m2) in therapy combinations with the chemotherapeutic agents 5-FU, Oxaliplatin +/- bevcizumab, and Irinotecan.

When the selected phase 2 dose is determined, 40 additional patients, will be included in the study in order to acquire more data on the safety and tolerability of Modufolin at this dose level. Twenty (20) of these additional patients will be treated in with Oxaliplatin, 20 with Irinotecan.

ELIGIBILITY:
Inclusion Criteria:

Advanced metastatic colorectal (Stage IV) cancer verified by biopsy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 105 (Actual)
Dates: Start 2014-09 (Actual); Primary Completion 2020-01-30 (Actual); Study Completion 2020-01-30 (Actual)

PRIMARY OUTCOMES:
Frequency and severity of dose limiting toxicity (DLT) or other Adverse Events (AE) | The patients will be followed during 4 cycles of treatment (8 weeks).
  Primary safety variables will consist of monitoring and recording of DLTs and any significant AE that have led to adjustments in the therapy administration.

CONTACTS AND LOCATIONS:
Overall Officials: Göran Carlsson, MD, Principal Investigator — Sahlgrenska University Hospital
Locations (10):
- Odense University Hospital, Odense, Denmark
- Greece (5):
  - 251 General Airforce Hospital, Athens
  - Medical School University of Athens, Aretaieio Hospital, Athens
  - Metropolitan General Hospital, Athens
  - University Genral Hospital Attikon, Athens
  - University General Hospital of Heraklion, Irakleio
- Norway (2):
  - Oslo University Hospital - Radiumhospitalet, Oslo
  - Oslo University Hospital - Ullevål, Oslo
- Sweden (2):
  - Sahlgrenska University Hospital, Gothenburg
  - Skaraborg hospital, Skövde

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Carlsson G, Koumarianou A, Guren TK, Haux J, Katsaounis P, Kentepozidis N, Pfeiffer P, Braendengen M, Mavroudis D, Taflin H, Skintemo L, Tell R, Papadimitriou C. A phase I/II study of arfolitixorin and 5-fluorouracil in combination with oxaliplatin (plus or minus bevacizumab) or irinotecan in metastatic colorectal cancer. ESMO Open. 2022 Oct;7(5):100589. doi: 10.1016/j.esmoop.2022.100589. Epub 2022 Sep 29. PMID 36183444
- [Derived] Taflin H, Odin E, Carlsson G, Tell R, Gustavsson B, Wettergren Y. Plasma deoxyuridine as a surrogate marker for toxicity and early clinical response in patients with metastatic colorectal cancer after 5-FU-based therapy in combination with arfolitixorin. Cancer Chemother Pharmacol. 2021 Jan;87(1):31-41. doi: 10.1007/s00280-020-04173-2. Epub 2020 Oct 24. PMID 33099678